CLINICAL TRIAL: NCT06667544
Title: A Phase 1/2, First-in-Human, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of RNK08954 in Patients With Advanced Solid Tumors With a KRAS G12D Mutation TRIAD1 (Trial of RNK08954 In KRAS G12D Mutation)
Brief Title: A Study of RNK08954 in Subjects With Advanced Solid Tumors With KRAS ((Kirsten Rat Sarcoma) G12D Mutation
Acronym: TRIAD1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ranok Therapeutics (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ranok Therapuetics Co. Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNK08954-01
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: KRAS G12D Mutation

STUDY DESIGN:
Intervention Model Description: PK-guided single-patient cohort followed by, A U-BOIN (Utility-based Bayesian Optimal Interval) design, with an incorporated Accelerated Titration (AT) step in the first dose level and then will enroll a minimum of 3 patients per dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RNK08954 (Experimental): Dose-escalation of RNK08954 oral dose therapy once daily.
  Interventions: Drug: RNK08954-01

INTERVENTIONS:
Drug: RNK08954-01 — Once daily oral treatment for a 3 week cycle

SUMMARY:
This is a first in human (FIH), Phase 1/2 open-label multi-center, dose escalation and expansion study to evaluate the safety, tolerability and pharmacokinetics of RNK08954 to determine the optimal dose and recommended dose for expansion and evaluate clinical activity in patients with advanced solid tumors with KRAS G12D mutation.

This is a 2-part study: dose exploration/indication expansion and dose optimization ( to identify a dose that preserves clinical benefit with optimal tolerability).

DETAILED DESCRIPTION:
In Phase 1a, enrolled subjects will receive oral RNK08954 daily after one subject completes a Lead-in Pharmacokinetic (PK) guided single-patient cohort. The dose escalation cohorts will start with one patient per cohort for the first dose levels, then will enroll a minimum of 3 patients per dose level. Five dose levels will be explored and a total of 42 patients are projected for enrollment.

Phase 1b- Multiple Indications Cohorts will open once the optimal dose has been determined in Phase 1a, and will consist of 3 cohorts including colorectal cancer, pancreatic adenocarcinoma and other indications. Approximately 20 patients will be assigned to each of the 3 cohorts for a total of 60 patients. All enrollment will be concurrent. Enrolled subjects will receive oral RNK08954 daily.

Phase 2 Dose Optimization Study will enroll subjects who will receive two different doses of oral RNK08954 daily to compare two different doses and further characterize the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older.
2. Must have pathologically documented locally advanced or metastatic malignancy harboring KRAS G12D mutations identified through deoxyribonucleic acid (DNA) sequencing of tumor tissues or circulating deoxyribonucleic acid (ctDNA) performed locally.
3. Must have received prior standard therapy appropriate for their tumor type, or in the opinion of the investigator, would be unlikely to derive further clinically meaningful benefit from appropriate standard of care therapy.
4. Must have measurable lesion(s) per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 by Computed tomography (CT) scan with contrast (magnetic resonance imaging (MRI), if the patient is allergic to contrast media).

   * Measurable disease may be in the field of prior irradiation; however, at least 3 weeks must have elapsed between the completion of radiation therapy and the baseline scan documenting disease status.
   * Bone disease is considered radiologically measurable only if there is at least a 50% lytic component.

   NOTE: Bone disease consisting of only blastic lesion is not considered measurable.

   NOTE: in Phase 1a, patients must have measurable or evaluable disease.
5. Archival or fresh tumor tissue must be available for evaluating relevant biomarkers. Formalin-fixed paraffin-embedded (FFPE)block preferred, or a minimum of 3 unstained FFPE slides of one archived block is required.

   NOTE: cytology samples from fine needle aspirates or brushing biopsies are not sufficient.

   NOTE: Phase 1a and 1b: Patients are additionally encouraged to undergo pre-treatment tumor biopsy.
6. Must have adequate performance status, Appendix D.

   o Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0, or 1.
7. Must be able to take oral medications and willing to record daily adherence to the investigational product.
8. Must have adequate laboratory parameters at baseline:

   * Absolute neutrophil count ≥ 1.2 x 109/L.
   * Hemoglobin greater than or equal to (≥) 9 g/dL.
   * Platelet count ≥ 75 x 109/L.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to (≤) 2.5 x upper limit of normal (ULN) (≤ 5 x ULN in presence of liver metastases).
   * Total bilirubin ≤ 1.5 x institutional ULN [less than (<) 2.5 x ULN for patients with documented Gilbert's syndrome or < 3.0 x ULN for patients for whom the indirect bilirubin level suggests an extrahepatic source of elevation].
   * Calculated creatinine clearance greater than (>) 60 mL/min. Actual body weight should be used for calculating creatinine clearance (e.g. using the Cockcroft-Gault formula).

   For patients with a Body Mass Index (BMI) > 30 Kg/m2, lean body weight should be used instead.
   * Acceptable coagulation parameters: Fibrinogen ≥ 1.5 g/dL, or partial thromboplastin time (PTT) ≤ 1.5 X institutional ULN, or international normalized ratio (INR) < 1.5 X institutional ULN or within target range if a patient is on prophylactic anti-coagulant therapy.
   * Serum albumin ≥ 3.0 g/dL.
9. Must have life expectancy of > 12 weeks according to the Investigator's clinical judgment.
10. Females of childbearing potential must have a negative pregnancy test at screening and additional pregnancy test prior to first dose.

    NOTE: Positive pregnancy test may occur in approximately 10% of cancer patients, who are otherwise postmenopausal. This is due to Human Chorionic Gonadotrophin (HCG) secreted by some tumor types such as ovarian or colorectal cancer (CRC), even in postmenopausal women. A quantitative test should be performed in patients with a positive serum pregnancy test, otherwise thought to be postmenopausal.
11. Males and females of childbearing potential must agree to use a highly effective method of contraception during treatment and for at least 6 months after the last dose of study treatment. These include, but not limited to:

    o Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (i.e. intravaginal or transdermal).
    * Progestogen-only hormonal contraception associated with inhibition of ovulation (i.e. injectable or implantable).
    * Intrauterine device.
    * Bilateral tubal occlusion.
    * Vasectomized partner.
    * Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments) is intended. The true abstinence is when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g. calendar, ovulation, symptom-thermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

    NOTE: A patient is not considered in childbearing potential if any of the following criteria is met:
    * has had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
    * Age ≥ to 60 years and is amenorrhoeic.
    * Age < 60 years and has been amenorrhoeic for ≥12 months (including no irregular menses or spotting) in the absence of any medication which induces a menopausal state and has ovarian failure as indicated by serum estradiol and follicle-stimulating hormone levels.

    NOTE: Male patients will be advised to arrange for the freezing of sperm samples prior to the start of the study, and not to donate sperm until 6 months after discontinuation of study treatment.
12. Must be able to understand and comply with the conditions of the protocol and must have read and understood the consent form and provided written informed consent.

    Food Effect Assessment- Specific Inclusion Criteria
13. Must be able to eat a standardized high-fat, high-caloric meal within 30 minutes.
14. Must be able to fast for a minimum of 10 hours. Phase 1b and Phase 2 Specific inclusion criteria
15. Patient must have received at least one but no more than two prior lines of systemic cytotoxic chemotherapy in locally advanced or metastatic setting.
16. The status of KRAS G12D mutations will be performed in a central laboratory chosen by the Sponsor.

Exclusion Criteria:

A patient is not eligible to participate in the study if any of the following criteria are met:

1. Concurrent anticancer therapy [chemotherapy, monoclonal antibodies, targeted therapy, hormonal therapy or investigational agents] within the lesser of 28 days or 5 half-lives before study Day 1.

   NOTE: Patient must agree not to participate in any other interventional clinical studies during their participation in this trial while on study treatment.

   NOTE: patients receiving hormonal ablation therapy for breast cancer or hormone refractory prostate cancer are allowed.

   NOTE: Patients taking part in surveys or observational studies are eligible to participate in this study.
2. Significant acute decline in clinical status including:

   -Decline in ECOG PS to >1 between baseline visit and within 72 hours prior to starting study treatment.

   -Weight loss of ≥10% during screening.
3. Presence of active or symptomatic untreated central nervous system (CNS) metastases.

   NOTE: Patients with asymptomatic or stable CNS metastases are eligible, provided that the CNS metastases are radiologically and clinically stable for at least 2 weeks prior to enrollment, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
4. Unresolved toxicities from prior anticancer therapy, defined as not having resolved according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade ≤ 1, or to levels dictated in the eligibility criteria, with the exception of alopecia.

   NOTE: Grade 2 or 3 toxicities from prior anticancer therapy that are considered irreversible (present and stable for >6 months) may be allowed if they are not otherwise described in the exclusion criteria and after a consultation between the Medical Monitor and the Investigator.
5. Prior radiotherapy to the only area of measurable disease, unless there is documented disease progression.

   NOTE: Patients must have completed treatment and recovered from all acute treatment-related toxicities prior to administration of the first dose of RNK08954.
6. Presence of gastrointestinal (GI) tract disease causing inability to take oral medication, such as malabsorption syndrome, requirement for intravenous alimentation, uncontrolled inflammatory GI disease, e.g. Crohn's disease or ulcerative colitis, or any other severe acute or chronic condition that may increase the risk of study participation including, e.g. history of abdominal fistula, GI perforation, peptic ulcer.
7. Current or history within 6 months prior to study enrollment of medically significant cardiovascular disease including symptomatic congestive heart failure > New York Heart Association (NYHA) Class II, unstable angina pectoris, clinically significant cardiac arrhythmia, or a history of long QT Syndrome (the heart's electrical activity as graphed on an electrocardiogram) or a family member with this condition.

   NOTE: patients with a marked baseline prolongation of QT/QTc (corrected) interval (e.g. repeated demonstration of a corrected QT (QTc) interval ≥ 470 mSec (one thousandth of a second) will be excluded. A consistent method of QTc calculation must be used for each patient's QTc measurements. QTcF (Fridericia's formula) is preferred.
8. Use of concomitant medications that have the potential to cause clinically relevant drug-drug interactions with RNK08954; including but not limited to:

   * All herbal medicines (e.g. St John's wort).
   * Use of strong inhibitors of Polymeric P-glycoprotein) P-gp within two weeks prior to Study Day 1.
   * Use of strong inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) within two weeks prior to Study Day 1.
   * Use of known 3A4, or C member 19 (2C19) sensitive substrates (with a narrow therapeutic window) within two weeks prior to Study Day 1.

   NOTE: other supplemental medicines, vitamins received by the patients within 3 weeks of the study enrollment will be reviewed and acknowledged or approved by the Investigator and the Sponsor Medical Monitor.
9. Pregnancy or breast-feeding or planning to breast feed during the study or within 6 months after study treatment.
10. Untreated human immunodeficiency virus (HIV). NOTE: Patients with a known history of HIV infection should have a cluster of differentiation 4 (CD4)+ thymus (T)-cell (CD4+) count ≥ 350 cells/mL to be eligible.
11. Active infection requiring systemic antibiotics, antiviral or antifungal treatment.

    NOTE: Patient must be medically stable, afebrile, and not taking antimicrobial treatment for ≤ 3 days prior to the first dose of study drug.
12. Known hepatitis B virus, or Hepatitis C virus:

    * Positive Hepatitis B Surface Antigen (Hep B sAg) (indicative of chronic Hepatitis B), positive Hepatitis total core antibody with negative Hep B sAg (suggestive of occult hepatitis B).
    * Detectable Hepatitis C virus (HCV) Ribonucleic acid (RNA) by Polymerase chain reaction (PCR) (indicative of active Hepatitis C), or positive Hepatitis C Antibody (Hep C Ab).

    NOTE: testing at screening is not required unless clinically indicated by the Investigator.

    NOTE: Patients with a history of hepatitis B or C are allowed if hepatitis B virus (HBV )DNA or hepatitis C virus (HCV) RNA are undetectable.
13. Known hypersensitivity to any of the components of the study drug.
14. Other conditions, psychiatric illness/social situations or any other serious uncontrolled medical disorders in the opinion of the Investigator that would limit compliance with study requirements.

Phase 1b and Phase 2 Specific exclusion criteria 15. History of other malignancies except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated by surgery alone or surgery plus radiotherapy with no evidence of disease for >2 years.

16. Prior treatment with KRAS G12D or Pan KRAS inhibitor.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs). | 12-15 months
  To evaluate the safety and tolerability of RNK08954 in adult patients with KRAS G12D mutant solid tumors in approximately 42 subjects
Optimal Biological Dose (OBD). | 12-15 months
  To determine the Recommended Dose for Expansion (RDE) of RNK08954 monotherapy in adult patients with KRAS G12D mutant solid tumors.

SECONDARY OUTCOMES:
Dose limiting toxicities (DLT) | 12-15 months
  To Determine Maximum Tolerated Dose (MTD) of RNK08954 monotherapy in adult patients with KRAS G12D mutant solid tumors
Objective response rate (ORR) | 12-15 months
  To determine the clinical activity of RNK08954 as monotherapy
Overall survival (OS), 1-year survival rate. | 12-15 months
  To determine the clinical activity of RNK08954 as monotherapy
.Evaluate Area under the plasma concentration (AUC0-72) in the fasted and fed states. | 12-15 months
  To evaluate the effect of food on the exposure of RNK08954

CONTACTS AND LOCATIONS:
Overall Officials: Zhengbo Song, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (6):
- China (6):
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No